CLINICAL TRIAL: NCT02568865
Title: Non-Invasive Physiologic Sensors to Assess Depression
Brief Title: Noninvasive Physiologic Sensors to Assess Depression
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, Director, Depression Clinical and Research Program, Massachusetts General Hospital
Other Study IDs: 2015P001913
Record Dates: First submitted 2015-09-14; First posted 2015-10-06 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Major Depressive Disorder
  Interventions: Other: Physiological Sensors; Other: Sleep Monitoring Device; Other: Vocal Monitoring; Other: Mobile Phone
- Healthy Volunteers
  Interventions: Other: Physiological Sensors; Other: Sleep Monitoring Device; Other: Vocal Monitoring; Other: Mobile Phone

INTERVENTIONS:
Other: Physiological Sensors — Wearable biosensors can play an important role in depression diagnosis. For this study, we will use a cost-effective, unobtrusive, and non-stigmatizing sensor to monitor physiological signals (including heart rate (HR), heart rate variability (HRV), electrodermal activity (EDA), physical activity, and temperature).
Other: Sleep Monitoring Device — The X4 Device is an internally battery powered FDA-classified Type BF device used for configurable acquisition of physiological signals via EEG.
Other: Vocal Monitoring — The participants will be provided with a phone app to leave audio diary recordings.
Other: Mobile Phone — A mobile phone and tablet will be used for various purposes, including, recording of socialization, location, and activity patterns of participants and to collect emotional information based on interactive surveys, as well as for forwarding sleep and physiological sensor measurements to a secure server.

SUMMARY:
This project aims to use sensors to monitor physiological signals, sleep patterns, vocal characteristics, activity, location and phone usage in study patients with depression who are receiving standard treatment (compared with healthy controls).

ELIGIBILITY:
Inclusion Criteria:

Patients with Depression (n=40):

1. Adults (ages 18-75),
2. Able to read, understand, and provide written informed consent in English,
3. Meet criteria for a primary psychiatric diagnosis of major depressive disorder for ≥ 4 weeks, according to the M.I.N.I (Mini International Neuropsychiatric Interview),
4. Hamilton Depression Rating Scale (HDRS) total score ≥ 18,
5. Engaged in or willing to be referred for clinical care for depression treatment as usual (antidepressants and/or psychotherapy),
6. Must have measurable skin conductance/electrodermal activity (as assessed at the screening visit),
7. Must own a working Android smartphone (Android 2.3+) and use it regularly,
8. Must own a windows PC (or tablet) or a Mac computer (or laptop),
9. Must have access to Internet service every day.

Healthy Controls (n=10):

1. Adults (ages 18-75),
2. Able to read, understand, and provide written informed consent in English,
3. Not meet criteria for past or current psychiatric illness, excluding specific phobias, as measured by the M.I.N.I.,
4. Not have a first-degree relative with known major psychiatric illness including Major Depressive Disorder, Bipolar Disorder, Psychotic Disorder or Substance Use Disorder,
5. Must have measurable skin conductance/electrodermal activity (as assessed at the screening visit),
6. Must own a working Android smartphone (Android 2.3+) and use it regularly,
7. Must own a windows PC (or tablet) or a Mac computer (or laptop),
8. Must have access to Internet service every day.

Exclusion Criteria (for all subjects):

1. Active drug or alcohol use disorder in the past 3 months,
2. History of psychosis,
3. History of mania or hypomania,
4. Epilepsy or history of seizures,
5. Untreated hypothyroidism,
6. Unstable medical disease,
7. Cognitive impairment that would impede adherence to study procedures,
8. Acute suicide or homicide risk,
9. Current treatment with electroconvulsive therapy, vagal nerve stimulation therapy, deep brain stimulation, transcranial magnetic stimulation therapy, or phototherapy,
10. Concurrent participation in other research studies,
11. Cannot comprehend or communicate in English,
12. Lack of working smartphone or lack of daily access to Internet service,
13. Inability to measure skin conductance/electrodermal activity (as assessed at the screening visit), and
14. Inability or unwilling to, at minimum, wear the physiological sensor (E4) bands, fill out the surveys, and record a weekly diary.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult outpatients with a current major depressive episode (n=40) and healthy adult controls (n=10).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Physiologic Biorhythms (heart rate) | 8 weeks
  We will measure the heart rate at baseline and during the treatment period. We will compare the corresponding patterns in patients with depression, as well as in healthy controls.
Phone Usage | 8 weeks
  We will measure the cell-phone usage (in the form of texts, web browsing, and phone calls) at the beginning of the study and during the treatment period. We will compare the corresponding phone usage patterns in patients with depression, as well as in healthy controls.
Voice Characteristics | 8 weeks
  We will measure the voice characteristics (via reading a 30-second script as part of an audio diary) at the beginning of the study and during the treatment period. We will compare the corresponding voice characteristics in patients with depression, as well as in healthy controls.
Physiologic Biorhythms (Skin conductance) | 8 weeks
  We will measure the skin conductance at baseline and during the treatment period. We will compare the corresponding patterns in patients with depression, as well as in healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States